CLINICAL TRIAL: NCT00003658
Title: A Phase I-II Study of Pentostatin With Cyclophosphamide for Previously Treated Patients With Intermediate and High-Risk Chronic Lymphocytic Leukemia
Brief Title: Pentostatin, Cyclophosphamide, and Rituximab in Treating Patients With Chronic Lymphocytic Leukemia or Other B-cell Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-083; CDR0000066751 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1482
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenström macroglobulinemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — Filgrastim; Rituximab; Cyclophosphamide; Pentostatin

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: pentostatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining pentostatin, cyclophosphamide, and rituximab in treating patients who have chronic lymphocytic leukemia or other B-cell cancers that have been treated previously.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose of cyclophosphamide, with filgrastim (G-CSF) support, that can be safely administered with pentostatin and rituximab in patients with previously treated intermediate- or high-risk chronic lymphocytic leukemia or other low-grade B-cell malignancies. (Phase I closed to accrual effective 11/27/2001.)
* Characterize the toxicity of this regimen in these patients.
* Determine the incidence of response in these patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of cyclophosphamide (CTX).

* Phase I: Patients receive CTX IV followed by pentostatin IV on day 1 of course 1. Patients also receive filgrastim (G-CSF) subcutaneously once daily beginning on day 3 and continuing until blood counts recover. During the second and subsequent courses, patients receive CTX IV, pentostatin IV, and rituximab IV on day 1. Patients also receive G-CSF as in course 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with at least a partial response after the third course receive an additional 3 courses.

Cohorts of 3-6 patients receive escalating doses of CTX until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

(Phase I closed to accrual effective 11/27/2001.)

* Phase II: Patients receive CTX at the recommended phase II dose and treatment as above.

Patients are followed at least every 3 months for 1 year and then periodically thereafter.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for the phase I portion of this study. (Phase I closed to accrual effective 11/27/2001.) A total of 14-30 patients will be accrued for the phase II portion of this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Intermediate- or high-risk chronic lymphocytic leukemia (CLL) as defined by the three-stage Rai system

  * Rai intermediate disease must be active disease (including weight loss, fatigue, fevers, evidence of progressive marrow failure, splenomegaly, progressive lymphadenopathy, and progressive lymphocytosis with a rapid doubling time)
* Other low-grade B-cell neoplasms, including small lymphocytic lymphoma (and its variants), Waldenstrom's macroglobulinemia, and follicular lymphoma allowed
* Autoimmune hemolytic anemia or autoimmune thrombocytopenia allowed regardless of disease stage
* B-cells demonstrated by immunophenotypic (or immunohistochemical) analysis of the malignant lymphocytes
* Must be previously treated
* For CLL, absolute lymphocytosis in the blood at least 5,000 lymphocytes/mm^3 OR
* Bone marrow lymphocytosis at least 30% of all nucleated cells
* No Rai intermediate-risk disease that meets the criteria of Montserrat "smoldering leukemia" NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 4 weeks

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No active infections requiring systemic antibiotics
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy
* Concurrent intravenous immunoglobulin allowed
* Concurrent epoetin alfa allowed

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent prednisone therapy allowed as long as dose is stable or decreasing over the past 4 weeks
* No increase in prednisone therapy while on study

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1998-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Adam Weiss, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Lamanna N, Kalaycio M, Maslak P, Jurcic JG, Heaney M, Brentjens R, Zelenetz AD, Horgan D, Gencarelli A, Panageas KS, Scheinberg DA, Weiss MA. Pentostatin, cyclophosphamide, and rituximab is an active, well-tolerated regimen for patients with previously treated chronic lymphocytic leukemia. J Clin Oncol. 2006 Apr 1;24(10):1575-81. doi: 10.1200/JCO.2005.04.3836. Epub 2006 Mar 6. PMID 16520464
- [Result] Weiss MA, Maslak PG, Jurcic JG, Scheinberg DA, Aliff TB, Lamanna N, Frankel SR, Kossman SE, Horgan D. Pentostatin and cyclophosphamide: an effective new regimen in previously treated patients with chronic lymphocytic leukemia. J Clin Oncol. 2003 Apr 1;21(7):1278-84. doi: 10.1200/JCO.2003.08.100. PMID 12663715